CLINICAL TRIAL: NCT03004014
Title: Comparison Between Natural Sleep Endoscopy and Drug-induced Sleep Endoscopy Among Obstructive Sleep Apnea Subjects Referred for Surgical Treatment
Brief Title: Natural Sleep and Drug-induced Sleep Endoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pedro Rodrigues Genta (Other)
Responsible Party: Sponsor-Investigator, Pedro Rodrigues Genta, Principal Investigator, University of Sao Paulo General Hospital
Organization: University of Sao Paulo General Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: 13900
Record Dates: First submitted 2016-08-04; First posted 2016-12-28 (Estimated); Last update posted 2018-07-31 (Actual); Status verified 2018-07

CONDITIONS: Obstructive Sleep Apnea
Keywords: sleep endoscopy; sedation
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Natural Sleep (No Intervention): OSA subjects referred for surgical treatment will evaluated endoscopically during natural sleep
- Propofol Induced Sleep (Other): Sleep endoscopy during propofol induced sleep
  OSA subjects referred for surgical treatment will be evaluated endoscopically during propofol induced sleep
  Interventions: Other: Sleep endoscopy during propofol induced sleep

INTERVENTIONS:
Other: Sleep endoscopy during propofol induced sleep — It will be performed a sleep endoscopy during drug induced sleep endoscopy
  Arms: Propofol Induced Sleep

SUMMARY:
Drug induced sleep endoscopy (DISE) has been performed worldwide since 1991 to determine the site and configuration of upper airway obstruction in patients with obstructive sleep apnea (OSA). However, there are no studies comparing DISE to sleep endoscopy during natural sleep. Objectives: To compare DISE to natural sleep endoscopy in OSA patients referred for surgical treatment.

Methods: OSA patients referred to surgical treatment (lateral pharyngoplasty) will be enrolled in this study. Natural sleep endoscopy will be performed at the sleep lab during the night. Propofol induced sleep will be performed at the operating room before surgery. The VOTE (velum, oropharyngeal lateral walls, tongue base and epiglottis) classification will be used to compare site and configuration of collapse between studies. Peak inspiratory flow will also be compared between studies.

DETAILED DESCRIPTION:
Drug induced sleep endoscopy (DISE) has been performed worldwide since 1991 to determine the site and configuration of upper airway obstruction in patients with obstructive sleep apnea. However, there are no studies comparing DISE to sleep endoscopy during natural sleep. Objective: to compare natural sleep endoscopy to drug induced sleep with propofol.

The study population will include 28 patients who are candidates to surgical treatment.

Methods Detailed clinical history and physical examination will be performed before natural sleep endoscopy. A 2-hour fast will be required. During both natural sleep and propofol-induced sleep, pharyngeal pressure will be measured using a pressure-tipped catheter (model TC-500XG; Millar).The nasopharynx will be numbed with xylocaine (10%) and oxymetazoline (0.05%), the catheter will be passed through a nasal mask into one nostril, and placed at the tongue base as confirmed by visual inspection of the oropharynx.A 2.8mm pediatric bronchoscope (Olympus) will be passed through the mask and into the other nostril. A nasal mask will be fitted and a heated pneumotachograph with differential pressure transducer connected to the mask will quantify airflow. The endoscope will be located at velopharynx, lateral wall of the pharynx and 2 cm above tongue and epiglottis.The VOTE Endoscopic Classification will be used to describe site and configuration of pharyngeal collapse in each study. The study will be scored by two experienced investigators, blind to the patient identification and type of study (natural sleep or drug-induced). Propofol-induced sleep will be performed at the operating room before surgery.

ELIGIBILITY:
Inclusion Criteria:

* BMI less than 35kg/m2
* Apnea-hypopnea index > 5 events/hour of sleep
* Clinical indication of surgical treatment for sleep apnea

Exclusion Criteria:

* Severe or decompensated cardiac or respiratory diseases
* Previous pharyngeal surgery
* Tonsils grade III or IV
* Other sleep disturbance (parasomnias, primary insomnia, narcolepsy)
* Sedative medication use (opioids, benzodiazepines and muscle relaxants)
* Uncontrolled diabetes or hyperthyroidism

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2015-01; Primary Completion 2017-12 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
The VOTE Endoscopic Classification | Immediately, during the procedure
  Comparison of site and configuration of endoscopy findings between the natural and drug-induced sleep endoscopy. The VOTE Endoscopic Classification describes the patterns and the degree of obstruction during sleep endoscopy.

SECONDARY OUTCOMES:
Peak inspiratory flow | Immediately, during the procedure
  Peak inspiratory flow measured during both natural and drug-induced sleep endoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Pedro R Genta, Post Doc, Principal Investigator — Sleep Laboratoy, Heart Institute
Locations (1):
- Sleep Laboratory, Heart Institute, Pulmonary Division, Hospital das Clínicas da Universidade de São Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Ordones AB, Grad GF, Cahali MB, Lorenzi-Filho G, Sennes LU, Genta PR. Comparison of upper airway obstruction during zolpidem-induced sleep and propofol-induced sleep in patients with obstructive sleep apnea: a pilot study. J Clin Sleep Med. 2020 May 15;16(5):725-732. doi: 10.5664/jcsm.8334. Epub 2020 Feb 7. PMID 32029070